CLINICAL TRIAL: NCT02215824
Title: A Randomised, Double-blind, Placebo-controlled, Dose Escalation Study to Investigate Safety, Pharmacokinetics and Pharmacodynamics of Different Doses (0.2, 0.6, 2.0, 6.0, and 20.0 μg/hr) of BIWH 3 Administered for 6 Hours in Patients With Chronic Critical Limb Ischaemia (CLI, Fontaine Class III or IV). COINART-1 Trial (First COllateral INto ARTery Trial)
Brief Title: Investigation of Safety, Pharmacokinetics and Pharmacodynamics of Different Doses of BIWH 3 in Patients With Chronic Critical Limb Ischaemia
Acronym: COINART-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1181.1
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

ARMS (2):
- BIWH 3 (Experimental): in escalating doses
  Interventions: Drug: BIWH 3
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIWH 3
  Arms: BIWH 3
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary aim of this trial was to investigate the safety of a 6 hour intraarterial infusion of BIWH 3 (pyro-Glu-rhMCP-1) in patients with severe peripheral arterial occlusive disease (PAOD) and chronic Critical Limb Ischaemia (Fontaine class III or IV).

ELIGIBILITY:
Inclusion:

* Patient must have severe PAOD with Chronic Critical Limb Ischaemia, Fontaine class III (ischaemic pain at rest) or IV (tissue ulceration or gangrene) due to atherosclerotic disease
* Patient must be >= 18 years of age
* Patient must give written informed consent
* Patient must have a life expectancy of at least six months

Exclusion:

* Transient ischaemic attack (TIA), cerebral vascular accident (CVA), myocardial infarction (MI) or episode of unstable angina within the past two months
* Ophthalmologic conditions: moderate to severe nonproliferative retinopathy, proliferative retinopathy, age related maculopathy with choroidal neovascularisation, macular edema, intraocular surgery within the previous 6 months, retinal vein occlusion
* Presence of a clinically significant disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the result of the study or the patient's ability to participate in the study
* ECG results outside of the reference range of clinical relevance including, but not limited to QTcB > 480 msec, PR interval > 240 msec, QRS interval > 140 msec
* History of malignant disease, or a positive result on any of the required cancer screening tests, unless a definitive subsequent evaluation for cancer is determined to be negative
* Patients at increased risk of colorectal cancer, including any of the following (1) colorectal cancer pr polyps in a first-degree relative younger than 60 or in two first-degree relatives of any age, (2) family history of familial adenomatous polyposis or hereditary non-polyposis colon cancer, (3) history of adenomatous polyps, or (4) history of chronic inflammatory bowel disease (chronic ulcerative colitis or Crohn's disease)
* Abnormalities greater than two times the upper limit of normal in any of the following laboratory values at Visit 1: alanine-aminotransferase (ALT), aspartate-aminotransferase (AST), gamma-glutamyl transferase (GGT), alkaline phosphatase or lactic dehydrogenase (LDH); abnormalities greater than 1.5 times the upper limit of normal of total bilirubin or white blood cell count
* Any concurrent infectious disease requiring treatment
* Severe renal insufficiency (estimated creatinine clearance < 30 mL/min)
* Duffy antigen negative blood type with co-existing moderate to severe renal insufficiency (estimated creatinine clearance < 80 mL/min), to avoid potential risk of significant increase of monocyte chemoattractant protein-1 (MCP-1) levels
* Known glomerulonephritis, even if creatinine clearance is apparently normal
* Thrombocytopenia, i.e. platelet count <100,000 cells/μl at Visit 1
* History of drug or alcohol abuse within the past 2 two years or active drug or alcohol abuse, present alcohol intake more than three drinks per day
* Inability to comply with the protocol
* Treatment with an investigational drug within 30 days or 5 half-lives, whichever is greater before Visit 2
* Use of cilostazol if cilostazol therapy was started within 2 months prior to trial enrollment, or planned initiation of cilostazol therapy during the trial period. Patients who have been on cilostazol for > 2 months prior to enrollment may be enrolled
* Inability to discontinue the intake of coumadin until after completion of the treatment period. Patients who were on coumadin must have an international normalised ratio (INR) < 1.8 at Visit 2
* Previous enrollment in this trial
* Hypersensitivity or allergy to heparin, conventional angiographic contrast dye, or magnetic resonance angiography (MRA) contrast
* Inability to undergo MRA (e.g. heart pacemaker, artificial heart valve, implanted neurostimulator, intrauterine device (IUD), metallic ear implant, implanted port for delivering insulin, or other foreign or implanted or metallic objects such as bullet fragments, metal plates, pins, screws or staples, joint replacement, or penile implant)
* Know HIV-infection
* Unwillingness to take blood products
* Pregnancy (to be excluded by serum and urine beta-human chorionic gonadotropin-test in women of childbearing potential) or breast feeding
* Female of childbearing potential (not 12 months post-menopausal or surgically sterilized) not using one of the following methods of birth control: hormonal contraceptives, oral or injectable/implantable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2002-10; Primary Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 180 days after drug administration
Number of patients with clinically relevant changes in vital signs (heart rate, blood pressure, body temperature) | baseline, up to 180 days after drug administration
Number of patients with clinically relevant changes in laboratory evaluations | baseline, up to 180 days after drug administration
Number of patients with clinically relevant changes in 12- lead electrocardiogram (ECG) | baseline, up to 180 days after drug administration
Number of patients with clinically relevant changes in markers of inflammation | baseline, up to 180 days after drug administration
  measured by C-reactive Protein (CRP) and erythrocyte sedimentation rate (ESR)
Number of patients with clinically relevant changes in ophthalmic examinations | baseline, up to 180 days after drug administration
Number of patients with changes from baseline in progression of atherosclerosis | day 180
  measured by carotid duplex imaging
Number of patients with changes in local disease defined by degree of stenosis | up to 6 months post treatment
  assessed by magnetic resonance angiography
Number of patients with changes from baseline in result of cancer screening | day 180
Number of patients developing an antibody response to BIWH 3 | baseline, up to 180 days

SECONDARY OUTCOMES:
Changes in transcutaneous oxygen pressure (tcPO2) | baseline, up to 180 days after drug administration
Changes in lower extremity magnetic resonance angiography (MRA) | baseline, up to 180 days after drug administration
Changes in ankle brachial or toe brachial index | baseline, up to 180 days after drug administration
Occurence of amputations | up to 180 days after drug administration
Progression of ulcer healing | up to 180 days after drug administration
Changes from baseline on visual analogue scale assessment of pain at rest | up to 180 days after drug administration
BIWH 3 plasma concentration | up to 180 days after drug administration
Occurrence of Mac-1 positive staining monocytes | up to 180 days after drug administration